CLINICAL TRIAL: NCT06327646
Title: Non-inferiority Assessment of Maternal Adherence to Supplementation: a Trial on the Effects of MMS
Brief Title: Maternal Adherence to MMS in Nepal
Acronym: NAMASTE MMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Keller International (Other)
Collaborators: Eleanor Crook Foundation (Unknown); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Kenda Cunningham, Sr. Research Advisor, Helen Keller International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 66677
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Supplementation
Keywords: Multiple Micronutrient Supplementation; Iron Folic Acid; Pregnancy; Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IFA-180 (Blister) (Active Comparator)
  Interventions: Drug: Iron Folic Acid Blister
- MMS-180 (Blister) (Experimental)
  Interventions: Drug: Multiple Micronutrient Supplement Blister
- MMS-180 (Bottle) (Experimental)
  Interventions: Drug: Multiple Micronutrient Supplement Bottle

INTERVENTIONS:
Drug: Multiple Micronutrient Supplement Blister — MMS in a blister pack along with related job aids, counselling during ANC, etc.
  Arms: MMS-180 (Blister)
Drug: Multiple Micronutrient Supplement Bottle — MMS in bottles along with related job aids, counselling during ANC, etc.
  Arms: MMS-180 (Bottle)
Drug: Iron Folic Acid Blister — Standard of Care - IFA in a blister pack along with related job aids, counselling during ANC, etc.
  Arms: IFA-180 (Blister)

SUMMARY:
Although clinical studies highlight the value of MMS for pregnant and lactating women, implementation research studies are necessary to understand adherence and acceptability to the product and to uncover potential obstacles to implementation in specific contexts. For Nepal, it is crucial to establish whether adherence to MMS supplementation is non-inferior to the existing IFA supplementation for 180 tablets, which has a high (65%) adherence rate. It is also important to investigate how whether providing MMS in bottles (containing a substantial quantity, such as 90 count bottles twice during pregnancy) might impact ANC utilization, particularly in terms of ensuring that pregnant women attend at least eight ANC visits. Furthermore, assessment of MMS acceptability, including pill taste, smell, size, swallowability, side effects, benefits as well as aspects such as product labeling and packaging, among end users in Nepal, is needed to understand acceptability of MMS vs. IFA. Finally, implementation issues within the health system, including the need of trainings for healthcare workers' and, female community health volunteers (FCHVs)' training needs; and government stakeholders' interest and barriers;; community s Social and behavioral change communication needs, and issues around supply chain issues should be well-understood and documented to inform prior to scale-up to support a smooth transition of MMS. Thus, Helen Keller International, in collaboration with Nepal's Ministry of Health and Population (MoHP) and the Eleanor Crook Foundation (ECF), will conduct a set of four mixed-methods studies to generate evidence and insights that inform the development of an MMS supplementation strategy. This trial in one province of Nepal is the first study that will be complemented by one additional quantitative study and two qualitative studies to generate evidence on the topics mentioned.

DETAILED DESCRIPTION:
The primary and secondary research questions for the randomized controlled trial named "Non-inferiority Assessment of Maternal Adherence to Supplementation: A Trial of the Effects of MMS" (NAMASTE MMS) are detailed below:

Primary:

1. Is adherence to the full prescription of 180 MMS (-blister) during pregnancy non-inferior to adherence to the full prescription of 180 IFA-blister during pregnancy (arm 2 vs arm 1)?
2. Is adherence to the full prescription of 180 MMS (-bottle) during pregnancy non-inferior to adherence to the full prescription of 180 IFA-blister during pregnancy (arm 3 vs arm 1)?

Secondary:

1. Is the level of adherence to MMS-blister and MMS-bottle non-inferior to the level of adherence to IFA-blister at different points during pregnancy and lactation (i.e. 30 days, 90 days, and 45 days postpartum from start of supplementation) (arm 2 vs. arm 1 and arm 3 vs arm 1)?
2. Is there a difference in adherence to 180 MMS during pregnancy from blister packaging vs bottle packaging of MMS (arm 2 vs arm 3?
3. Is there a difference in adherence to ANC visits during pregnancy from blister packaging vs bottle packaging of MMS (arm 2 vs arm 3)?
4. What is the level of acceptability of IFA and MMS at different stages of pregnancy (i.e. 30 days, 90 days, 180 days, and 45 days postpartum) (arms 1, 2 and 3)?
5. What is the validity of women's recall of the amount of MMS/IFA received and of adherence to MMS/IFA compared to a gold standard?

This c-RCT will be conducted among pregnant women assigned to one of three trial arms (as described below in the section on interventional description). Data will be collected via in-person surveys at their home over a period of 12 months, including immediately following the 30-, 90-, delivery (180-) and 45-days post-partum (225-) day points post-enrollment at the pregnant woman's first antenatal care visit.

The c-RCT will be conducted in Lumbini Province of Nepal, which was purposely selected among the four provinces that cover all three agro-ecological regions in Nepal: mountains, hills, and the terai (plains) due to ease of implementation. The random sampling of health facilities (clusters) will be as proportional to the population as possible - i.e., 10% from mountains, 40% from hills, and 50% from terai. The required facilities (n=120) will be randomly selected and assigned to one of the three c-RCT arms using from the list of government health facilities (primary health care centers (PHCCs), and health posts (HPs) only).

A total of 120 health facilities will be randomly assigned to one of the three arms. Forty (40) health facilities will receive IFA in blister packs (current standard of care), 40 health facilities will receive MMS in blister packs, and 40 will receive MMS in bottles, and 40 will receive IFA in blister packs. These supplements will be distributed pregnant women who health workers identify as meeting study criteria and who provide verbal informed consent to be study participants. When a woman reports for antenatal care to a health facility that is part of the RCT, the health worker will identify whether she is at least 18 years and no more than 35 years of age. If so, the health work will start to complete an enrollment log (Annex 4) to document the pregnant woman's details such as name, phone number, other household members' phone number(s), and house location details. This enrollment log also includes the study eligibility criteria (specified below) to help the health worker know if the woman could participate in the study. If she is deemed eligible, the health worker will inform her about the study and the opportunity to participate including the research objectives and processes and share detailed information on supplementation including its timing, benefits, and potential side effects. The enrollment log thus will generate a record of all pregnant women considered for the study, those excluded by each of the study inclusion criteria, and the refusal rate for the study, based on the health worker's initial screening. The health worker will share information for each pregnant woman deemed to meet study inclusion criteria and who agrees to participate in the study with the enumerator assigned to that particular health facility, following a communication protocol (Annex 5). The enumerator will, in turn, enter the woman's data into his/her electronic enrolment log, visit the woman at her home to verify her eligibility based on the inclusion/exclusion criteria, and obtain her written informed consent. For those women who are confirmed to meet study inclusion/exclusion criteria and provide their written informed consent to participate, the enumerator will then administer the enrollment survey. Pregnant women enrolled in the study who continue to provide consent and remain in the study will be further interviewed at 30 and 90-days post enrollment, as well as at delivery (approximately 180-days post enrollment) and 45-days post-partum (approximately 225-days post enrollment)

The recruitment of pregnant women will continue in each health center facility on a rolling basis until the targeted number of women (2,640) total are enrolled. Recruitment is anticipated to take approximately 8 months, with quicker data collection in the plains given a larger number of pregnant women using services from these facilities and progressively slower data collection in the hills and mountains, due to lower population and in turn, less frequent pregnancies, and service usage . Additional delays in recruitment may occur due to adverse weather, greater clarity on pregnancy rates once enrollment starts, and other factors

ELIGIBILITY:
Inclusion criteria

To be eligible for the study, health facilities must meet four criteria:

1. public/government-run;
2. either a PHCC or HP at point of randomization;
3. implement the standard ANC package of care; and
4. have the top 50% average monthly caseloads for newly enrolled pregnant women (i.e. first ANC) for that specific agro-ecological zone (mountains - at least 5/month; hill - at least 8/month; and terai - at least 15/month) based on health management information system (HMIS) ANC data (July 16, 2021, to July 15, 2022).

To be eligible for the study, pregnant women must meet multiple criteria, at the point of enrollment:

1. be 18 - 35 completed years of age at health facility enrollment;
2. not planning to move/migrate for at least nine months after enrollment;
3. gestational age of at least 12 but not yet 14 weeks at time of health facility enrollment, estimated based on her last menstrual period (LMP) with exact calendar calculation confirmed during visit by enumerator;
4. pregnancy without any complications; not classified as severe anemic as well as high-risk pregnancy (i.e. not having the following conditions: diabetes, polycystic ovary syndrome, thyroid disease, kidney diseases, fibroids and severe mental/physical conditions that prevent study participation including unable to speak, attend ANC/PNC, take supplements or mental/cognitive impairment);
5. provides written informed consent to participate in the study; and
6. agrees to have enumerators visit the home at different data collection points.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2640 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-07-24 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pregnancy supplementation for 180 days: binary | Delivery
  Consumed at least 180 supplement tablets between study enrollment and delivery (MMS-blister vs IFA-blister; MMS-bottle vs. IFA blister)
Pregnancy supplementation for 180 days: continuous | Delivery
  Number of supplements consumed between study enrollment and delivery (MMS-blister vs IFA-blister; MMS-bottle vs. IFA blister)

SECONDARY OUTCOMES:
Full pregnancy supplementation: binary | Delivery
  Consumed at least the maximum number of supplement tablets eligible to consume between study enrollment and delivery (MMS-blister vs IFA-blister; MMS-bottle vs. IFA blister; MMS-bottle vs MMS-blister)
Full pregnancy supplementation: continuous | Delivery
  Number of supplements consumed between study enrollment and delivery (MMS-blister vs IFA-blister; MMS-bottle vs. IFA blister; MMS-bottle vs MMS-blister)
MMS supplementation for 180 days: Binary | Delivery
  Consumed at least 180 supplement tablets between study enrollment and delivery (MMS-blister vs MMS-bottle)
MMS supplementation for 180 days: continuous | Delivery
  Number of supplements consumed between study enrollment and delivery (MMS-blister vs. MMS-bottle)
Antenatal Care Utilization: binary | Delivery
  Received the recommended 8 ANC visits during pregnancy or not (MMS-blister vs MMS-bottle)
Antenatal Care Utilization: continuous | Delivery
  Number of ANC visits during pregnancy (MMS-blister vs. MMS-bottle)

OTHER OUTCOMES:
Pregnancy supplementation for 30 days: binary | 30 days post enrollment/pill eligibility
  Consumed at least 30 supplement tablets between study enrollment and 30 days later during pregnancy (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Pregnancy supplementation for 90 days: binary | 90 days post enrollment/pill eligibility
  Consumed at least 90 supplement tablets between study enrollment and 30 day follow-up visit during pregnancy (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Postpartum supplementation for 45 days: binary | 45 days post delivery
  Consumed at least 45 supplement tablets between delivery and 45 days later (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Pregnancy supplementation for 30 days: continuous | 30 days post enrollment/pill eligibility
  Number of supplements consumed between study enrollment and 30 days later (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Pregnancy supplementation for 90 days: continuous | 90 days post enrollment/pill eligibility
  Number of supplements consumed between study enrollment and 90 days later (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Postpartum supplementation for 45 days: continuous | 45 days post delivery
  Number of supplements consumed between delivery and 45 days later (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Supplement acceptability at 30-days: continuous | 30-days post enrollment
  Degree of acceptability of supplements measured as a sum (0-25) from a 5-point likert scale for each property (taste, color, swallowability, odor, and frequency) 30-days post-enrollment (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Supplement acceptability at 90-days: continuous | 90-days post enrollment
  Degree of acceptability of supplements measured as a sum (0-25) from a 5-point likert scale for each property (taste, color, swallowability, odor, and frequency) 90-days post-enrollment (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Supplement acceptability at 180-days: continuous | Delivery
  Degree of acceptability of supplements measured as a sum (0-25) from a 5-point likert scale for each property (taste, color, swallowability, odor, and frequency) after delivery (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)
Supplement acceptability at 45-days post-partum: continuous | 45-days post partum
  Degree of acceptability of supplements measured as a sum (0-25) from a 5-point likert scale for each property (taste, color, swallowability, odor, and frequency), at 45 days post-partum (IFA-blister vs MMS-blister; IFA-blister vs MMS-bottle; MMS-blister vs MMS-bottle)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Klemm, PhD, Study Director — Helen Keller International
Locations (119):
- Nepal (119):
  - Thada primary health care centre, Arghakhanchi, Lumbini Province
  - Khairapur health post, Bardiyā, Lumbini Province
  - Mathura haridwar health post, Bardiyā, Lumbini Province
  - Motipur health post, Bardiyā, Lumbini Province
  - Neulapur health Post, Bardiyā, Lumbini Province
  - Sanoshree health post, Bardiyā, Lumbini Province
  - Banakatawa primary health care centre, Bānke, Lumbini Province
  - Banakatti health post, Bānke, Lumbini Province
  - Basudevapur health post, Bānke, Lumbini Province
  - Bejapur health post, Bānke, Lumbini Province
  - Belahari health post, Bānke, Lumbini Province
  - Betahani health post, Bānke, Lumbini Province
  - Chisapani health post, Bānke, Lumbini Province
  - Ganapur health post, Bānke, Lumbini Province
  - Gangapur health post, Bānke, Lumbini Province
  - Hirminiya health post, Bānke, Lumbini Province
  - Holiya health post, Bānke, Lumbini Province
  - Indrapur health post, Bānke, Lumbini Province
  - Jaispur health post, Bānke, Lumbini Province
  - Kalaphata health post, Bānke, Lumbini Province
  - Kathkuiya health post, Bānke, Lumbini Province
  - Khajura primary health care centre, Bānke, Lumbini Province
  - Khaskarkado health post, Bānke, Lumbini Province
  - Laxmanpur primary health care centre, Bānke, Lumbini Province
  - Matahiya health post, Bānke, Lumbini Province
  - Narainapur health post, Bānke, Lumbini Province
  - Phattepur health post, Bānke, Lumbini Province
  - Puraina health post, Bānke, Lumbini Province
  - Puraini health post, Bānke, Lumbini Province
  - Rainyapur health post, Bānke, Lumbini Province
  - Saigaun Health Post, Bānke, Lumbini Province
  - Sonpur health post, Bānke, Lumbini Province
  - Titihiriya health post, Bānke, Lumbini Province
  - Udarapur health post, Bānke, Lumbini Province
  - Udayapur health post, Bānke, Lumbini Province
  - Gadhawa Health Post, Dāng, Lumbini Province
  - Hapur Health Post, Dāng, Lumbini Province
  - Lalmatiya Health Post, Dāng, Lumbini Province
  - Laxmipur Health Post, Dāng, Lumbini Province
  - Satbariya Health Post, Dāng, Lumbini Province
  - Shantinagar Health Post, Dāng, Lumbini Province
  - Sisahaniya Health Post, Dāng, Lumbini Province
  - Aama Health Post, Lumbini, Lumbini Province
  - Amuwa (Paschhim) Health Post, Lumbini, Lumbini Province
  - Asurena Health Post, Lumbini, Lumbini Province
  - Bhagawanpur Health Post, Lumbini, Lumbini Province
  - Bodabar Health Post, Lumbini, Lumbini Province
  - Chhapiya Health Post, Lumbini, Lumbini Province
  - Dhakadhai Primary Health Care Centre, Lumbini, Lumbini Province
  - Dhamauli Health Post, Lumbini, Lumbini Province
  - Ekala Health Post, Lumbini, Lumbini Province
  - Farena Health Post, Lumbini, Lumbini Province
  - Gajedi Health Post, Lumbini, Lumbini Province
  - Gonaha Health Post, Lumbini, Lumbini Province
  - Harnaiya Health Post, Lumbini, Lumbini Province
  - Jogada Health Post, Lumbini, Lumbini Province
  - Kamahariya Health Post, Lumbini, Lumbini Province
  - Karmahawa Health Post, Lumbini, Lumbini Province
  - Khudabagar Health Post, Lumbini, Lumbini Province
  - Lumbini Primary Health Care Centre, Lumbini, Lumbini Province
  - Majhagawa Health Post, Lumbini, Lumbini Province
  - Manmateriya Health Post, Lumbini, Lumbini Province
  - Masina Health Post, Lumbini, Lumbini Province
  - Motipur primary health care centre, Lumbini, Lumbini Province
  - Parroha Health Post, Lumbini, Lumbini Province
  - Roinihawa Health Post, Lumbini, Lumbini Province
  - Rudrapur Health Post, Lumbini, Lumbini Province
  - Sadi Health Post, Lumbini, Lumbini Province
  - Sakraun Pakadi Health Post, Lumbini, Lumbini Province
  - Semara Bazar Health Post, Lumbini, Lumbini Province
  - Shankarnagar Health Post, Lumbini, Lumbini Province
  - Sikatahan Health Post, Lumbini, Lumbini Province
  - Sipawa Health Post, Lumbini, Lumbini Province
  - Tenuhawa Health Post, Lumbini, Lumbini Province
  - Jagnnathpur Primary Health Care Centre, Nawalparasi West, Lumbini Province
  - Paklihawa health post, Nawalparasi West, Lumbini Province
  - Arkha Health Post, Pyūthān, Lumbini Province
  - Bangeshal Health Post, Pyūthān, Lumbini Province
  - Bhingri Primary Health Care Centre, Pyūthān, Lumbini Province
  - Damri Health Post, Pyūthān, Lumbini Province
  - Devisthan Health Post, Pyūthān, Lumbini Province
  - Okharkot Health Post, Pyūthān, Lumbini Province
  - Phopli Health Post, Pyūthān, Lumbini Province
  - Rajwara Health Post, Pyūthān, Lumbini Province
  - Sapdanda Health Post, Pyūthān, Lumbini Province
  - Syauliwang Health Post, Pyūthān, Lumbini Province
  - Aresh Health Post, Rolpa, Lumbini Province
  - Holeri Phc, Rolpa, Lumbini Province
  - Liwang Health Post, Rolpa, Lumbini Province
  - Nerpa Health Post, Rolpa, Lumbini Province
  - Nuwagaun Health Post, Rolpa, Lumbini Province
  - Pakhapani Health Post, Rolpa, Lumbini Province
  - Pang Health Post, Rolpa, Lumbini Province
  - Rank Health Post, Rolpa, Lumbini Province
  - Sirpa Health Post, Rolpa, Lumbini Province
  - Sulichaur Phc, Rolpa, Lumbini Province
  - Hukam Health Post, Rukum East, Lumbini Province
  - Kankri Health Post, Rukum East, Lumbini Province
  - Pokhara Health Post, Rukum East, Lumbini Province
  - Sisne Health Post, Rukum East, Lumbini Province
  - Taksera Health Post, Rukum East, Lumbini Province
  - Baskhor health post, Taulihawā, Lumbini Province
  - Birpur health post, Taulihawā, Lumbini Province
  - Chanai Health Post, Taulihawā, Lumbini Province
  - Ganeshpur health post, Taulihawā, Lumbini Province
  - Gugauli health post, Taulihawā, Lumbini Province
  - Haranampur primary health care centre, Taulihawā, Lumbini Province
  - Hariharpur healthpost, Taulihawā, Lumbini Province
  - Jahadi health post, Taulihawā, Lumbini Province
  - Krishnanagar health post, Taulihawā, Lumbini Province
  - Labani health post, Taulihawā, Lumbini Province
  - Maharajgunj primary health care centre, Taulihawā, Lumbini Province
  - Motipur health post, Taulihawā, Lumbini Province
  - Pakadi health post, Taulihawā, Lumbini Province
  - Patariya health post, Taulihawā, Lumbini Province
  - Pathardeiya health post, Taulihawā, Lumbini Province
  - Shivapur health post, Taulihawā, Lumbini Province
  - Sisawa health post, Taulihawā, Lumbini Province
  - Tilaurakot health post, Taulihawā, Lumbini Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cunningham K, Poudel S, Hoang MA, Gupta AS, Adhikari R, K C D, Mohan D, Rana Y, Lal BK, Thapa LB, Klemm R. Non-inferiority Assessment of Maternal Adherence to Supplements, a Trial on the Effects of Multiple Micronutrient Supplementation (NAMASTE-MMS) in Nepal: study protocol. Trials. 2025 Nov 13;26(1):502. doi: 10.1186/s13063-025-09031-1. PMID 41233886